## Effect of Monazite Sands in Patients with Osteoarthritis of the Knee

Ethical committee Protocol No: 3.160.891

Screening\_log

Documente date: May 03<sup>rd</sup>, 2019

## **SUBJECT SCREENING LOG**

| Study brief Title: | Effects of Sand Treatment on Osteoarthritis |
|--------------------|---------------------------------------------|
|--------------------|---------------------------------------------|

Official Title: Effect of Monazite Sands in Patients With Osteoarthritis of the Knee

Complete this log for every subject screened for inclusion in the study.

| Nº | Subject's name | Gender | Date of birth<br>(dd/mm/yyyy) | Date screened for eligibility (dd/mm/yyyy) | Subject<br>Eligible? <sup>1</sup> | If ineligible,<br>specify reason<br>for ineligibility | Investigator Initials<br>and Date |
|---|---|---|---|---|---|---|---|
| | МО | MOFO | FO | | ( ) Yes | | |
| | | I III O I O | | | ( ) No | | |
| | | MOFO | | | ( ) Yes | | |
| | | MOFO | | | ( ) No | | |
| | MOFO | MOFO | | | ( ) Yes | | |
| | | MOFO | | | ( ) No | | |
| | Мо го | M O F O | | | ( ) Yes | | |
| | | MOFO | | | ( ) No | 1 | |
| | MOFO | MOFO | | | ( ) Yes | | |
| | | MOFO | | | ( ) No | | |
| | MOFO | | | ( ) Yes | | | |
| | | | | ( ) No | | | |
| | МС | | 40.50 | | ( ) Yes | | |
| | | MOFO | | | ( ) No | | |

<sup>&</sup>lt;sup>1</sup>Legend: Inclusion Criteria: A) Joint pain related to daily activities; B) No morning joint stiffness greater than 30 minutes; C) Age between 30 and 95 years.

| Signature of the Principal Investigator: | Date: |
|------------------------------------------|-------|